CLINICAL TRIAL: NCT05823480
Title: A Multi-Center, Phase 1 Trial of Combining Anti-CD47 Antibody (Magrolimab) with Azacitidine As Post-Transplant Maintenance Therapy in Patients Who Underwent Allogeneic Hematopoietic Cell Transplantation for Treatment of High-Risk AML or MDS
Brief Title: Magrolimab in Combination with Azacitidine After Allogeneic HCTin Treating Patients with High-Risk AML or MDS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn -ctms
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22618; NCI-2023-02417 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22618 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-29; First posted 2023-04-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Stem Cell Transplantation; Azacitidine; Specimen Handling; Biopsy; magrolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (magrolimab, azacitidine) (Experimental): Patients undergo allo HCT per standard of care. Patients then receive magrolimab IV and azacitidine IV on study. Patients undergo ECHO or MUGA during screening and blood sample collection and bone marrow biopsy and aspirate throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography; Biological: Magrolimab; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allo HCT per standard of care
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspirate — Undergo bone marrow biopsy and aspirate
  Other Names: Human Bone Marrow Aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspirate
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Biological: Magrolimab — Given IV
  Other Names: Hu5F9-G4
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies how well the combination of magrolimab works with azacitidine after a donor stem cell transplant (allogeneic hematopoietic cell transplantation) in treating patients with high-risk acute myeloid leukemia or myelodysplastic syndrome. Magrolimab is a type of protein called an antibody. It is designed to target and block a protein called CD47. CD47 is present on cancer cells and is used by cancer cells to protect themselves from the body's immune system. Blocking CD47 with magrolimab may enable the body's immune system to find and destroy the cancer cells. Azacitidine is a chemotherapy drug that may prevent the return of acute myeloid leukemia or myelodysplastic syndrome by working in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Combining magrolimab and azacitidine may kill more cancer cells after allogeneic hematopoietic cell transplantation in patients with high-risk acute myeloid leukemia or myelodysplastic syndromes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Establish safety/feasibility and determine the recommended phase 2 dose (RP2D) of magrolimab in combination with a fixed dose of azacitidine when given as the maintenance therapy after reduced intensity conditioning allogeneic hematopoietic cell transplantation (HCT), in patients with high-risk acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

I. Estimate overall survival (OS), progression-free survival (PFS), cumulative incidence (CI) of relapse/progression, non-relapse mortality (NRM) at +100 days and 1-year post- maintenance therapy.

II. Estimate CI of acute graft-versus-host disease (GVHD) at 180 days post HCT, and chronic GVHD at one-year post-HCT.

III. Longitudinally characterize minimal residual disease (MRD+) status in patients receiving maintenance therapy.

IV. Feasibility of receiving magrolimab in combination with azacitidine as maintenance therapy in this patient population.

EXPLORATORY OBJECTIVES:

I. Characterize the presence and level of GVHD biomarkers and inflammatory cytokines in the first 100 days from the start of maintenance therapy.

II. Assess the possible correlation between chimerism kinetics by AlloHeme assay (per next generation sequencing [NGS] assay) and post-HCT relapse.

III. Describe kinetics of immune cell recovery and macrophage activation in the first-year post-HCT.

IV. Assess health related quality of life (QoL) and symptoms on days 1, 60, 90 and 180 after starting maintenance therapy.

OUTLINE: This is a dose-escalation study of magrolimab (MRD- patients only), followed by a dose-expansion study (MRD- and MRD+ patients).

Patients undergo allo HCT per standard of care. Patients then receive magrolimab intravenously (IV) and azacitidine IV on study. Patients undergo echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) during screening and blood sample collection and bone marrow biopsy and aspirate throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the patient and/or legally authorized representative (done within 30 days of HCT day 0).
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies.

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval.
* Age: 18-75 years old.
* Eastern Cooperative Oncology Group =< 2.
* Patients who are scheduled to undergo allogeneic HCT for AML with high-risk cytogenetics per European Leukemia Net (ELN) or MDS with International Prognostic Scoring System (IPSS) of intermediate 2 with poor risk cytogenetics or molecular markers. OR patients with MRD+ disease OR active disease with < 10% blast at the time of HCT.
* Patients who are scheduled to undergo their first or second HCT with reduced intensity conditioning regimen (any reduced intensity conditioning regimen per institutional standards is allowed), and regardless of GVHD prophylactic regimen.
* Allogeneic transplant regardless of donor type (matched, mismatched, haploidentical, etc.) or graft source (bone marrow or mobilized peripheral blood stem cells) are included.
* Pre-HCT exposure to anti-CD47 of hypomethylating agent (HMA) is allowed if no progression on therapy has been documented.
* Absolute neutrophil count (ANC) >= 1.5 (without the use of granulocyte-colony stimulating factor [GCSF] for last 2 weeks) (To be performed within 45 days prior to transplant unless otherwise stated).

  * NOTE: Transfusion (Red blood cells [RBC] or platelet) to achieve the above-mentioned counts is allowed.
* Platelet count >= 50K (To be performed within 45 days prior to transplant unless otherwise stated).

  * NOTE: Transfusion (RBC or platelet) to achieve the above-mentioned counts is allowed.
  * NOTE: Complete blood count (CBC) should be done within 2 weeks of day 1 of the protocol.
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease) (To be performed within 45 days prior to transplant unless otherwise stated).
* Aspartate transaminase (AST) =< 1.5X ULN (To be performed within 45 days prior to transplant unless otherwise stated).
* Alanine transaminase (ALT) =< 1.5 X ULN (To be performed within 45 days prior to transplant unless otherwise stated).
* Creatinine clearance of >= 60 mL/min per 24-hour urine test or the Cockcroft-Gault formula (To be performed within 45 days prior to transplant unless otherwise stated).
* Left ventricular ejection fraction (LVEF) >= 45% (To be performed within 45 days prior to transplant unless otherwise stated).
* If able to perform pulmonary function tests: forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusing capacity of the lung for carbon monoxide (DLCO) (diffusion capacity) >= 50% of predicted (corrected for hemoglobin). If unable to perform pulmonary function tests: oxygen (O2) saturation > 92% on room air. (To be performed within 45 days prior to transplant unless otherwise stated).
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. (To be performed within 45 days prior to transplant unless otherwise stated).
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Patient who underwent more than 2 allogeneic HCTs.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents (azacitidine or magrolimab).
* Females only: Pregnant or breastfeeding.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Known inherited or acquired bleeding disorders.
* Clinical suspicion of active central nervous system (CNS) involvement by MDS.
* Significant medical diseases or conditions, including but not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes, significant active infection and congestive heart failure (CHF) New York Heart Association (NYHA) class 3-4.
* Known or active hepatitis B or C infection or human immunodeficiency virus (HIV) infection in medical history.
* Prospective patients who, in the opinion of the principal investigator (PI), may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-09 (Estimated); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | The evaluation period of DLT is from starting study regimen (day + 1) to the first observation of DLT, or the end of the first cycle of Magrolimab maintenance (day +85) with a grace period of ±7days, whichever comes first. (Each cycle is 28 days)
  Dose limiting toxicities (DLT) are defined as any of the following events that are attributed at least possibly due to study regimen and occur from start of magrolimab (day +1) to the end of the first cycle of magrolimab maintenance (day +85 +/-7): Death, grade 3-4 non-hematological toxicities per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE 5.0), grade 4 hematological toxicities per NCI CTCAE 5.0 that last for more than 21 days. Will utilize the revised National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 for adverse events reporting.
Maximum tolerated dose (MTD) and recommended phase 2 dose (RPD) of magrolimab | The evaluation period of DLT is from starting study regimen (day + 1) to the first observation of DLT, or the end of the first cycle of Magrolimab maintenance (day +85) with a grace period of ±7days, whichever comes first. (Each cycle is 28 days)
  Will use the time-to-event Bayesian optimal interval (TITE-BOIN) design [1] to find the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D).

SECONDARY OUTCOMES:
Overall survival | Time period from start of protocol therapy to death regardless of cause, assessed up to 6 years
Progression free survival | Time from start of protocol therapy to relapse/progression, or death, whichever comes first, assessed up to 6 years
Cumulative incidence of relapse/progression (CIR) | Time of start of treatment to time of relapse/progression, assessed up to 6 years
  Will be estimated using the cumulative incidence.
Cumulative incidence of on-relapse mortality (NRM) | Time of start of treatment to non-disease related death, assessed up to 6 years
  Will be estimated using the cumulative incidence.
Cumulative incidence of acute graft versus host disease (aGvHD) of grades 2-4 and 3-4 | Time of start of treatment to first documented/biopsy proven acute GVHD onset date, at 180 days post transplant
  Will be assessed by documented or biopsy proven aGvHD and graded according to the Mount Sinai Acute GVHD International Consortium (MAGIC) grading. Will be estimated using the cumulative incidence curve.
Cumulative incidence of chronic graft versus host disease (cGvHD) | Time of start of treatment to first documented/biopsy proven chronic GVHD onset date, assessed at 1 year post transplant
  Will be assessed by documented or biopsy proven cGvHD and scored according to the National Institutes of Health (NIH) Consensus Staging. Disease relapse/progression or NRM is considered competing risk events. cGvHD will be censored at time of last follow-up if patients remain alive and free of relapse/progression. cGvHD will be estimated using the cumulative incidence curve.
Minimal residual disease | Assessed up to 6 years
  Will be assessed from bone marrow aspirates collected on days 30, 100, and 180 post HCT.
Completion of planned therapy | Assessed up to 6 years
  Feasibility is defined as ability to complete at least 30% of the planned therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr M Al Malki, MD, Principal Investigator — City of Hope Medical Center